CLINICAL TRIAL: NCT06260540
Title: Investigation of the Effect of Core Endurance Levels on Upper Extremity Function, Muscle Strength and Reaction Time in Healthy Young Adults
Brief Title: Core Endurance in Healthy Young Adults
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Other Study IDs: Core Endurance
Record Dates: First submitted 2024-02-06; First posted 2024-02-15 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Health Risk Behaviors
Keywords: core endurance; upper extremity function; muscle strength; reaction time
MeSH Terms: conditions — Health Risk Behaviors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to examine the effect of core endurance levels on upper extremity function, muscle strength and reaction time in healthy young adults. The "core" region functions as a connection point between the upper and lower extremities and enables the transfer of force from this region to the extremities. This region is a basic structure where the force required for all movements is generated and transmitted from the proximal segments to the distal segments. "Core" stabilization has a significant impact on limb functionality, and stabilization of the proximal segments is necessary to maintain the mobility and function of the distal segments. To establish a stable base during functional activities, the "core" muscles are activated before the upper and lower extremity muscles. This ensures force production and transfer of resulting forces, thus supporting the mobility of the distal segments. Increasing core stabilization increases force production in the extremities, and control of core strength, balance and movement maximizes upper and lower extremity functions. Any impairment in core stabilization reduces the quality of movement and increases the risk of injury to the upper extremity. Therefore, it has been stated that "core" stabilization has a significant effect on athletic performance and upper extremity functions. There are not enough studies in the literature investigating this effect in healthy young adults. Most existing studies focus on the role of core endurance on athlete performance.

The aim of this study is not only to investigate core endurance levels in healthy young adults but also to examine the effect of core endurance levels on upper extremity function, muscle strength and reaction time.

DETAILED DESCRIPTION:
The "core" region is depicted as a box or cylinder and includes the spine, hips, pelvis, proximal lower extremities, and abdominal structures. This region consists of the abdominals, gluteals, paraspinals, diaphragm, oblique abdominals, pelvic floor and hip girdle muscles. These muscles provide stabilization on the trunk and spine during movement or at rest. The "core" region consists of 29 pairs of muscles and these muscles are classified according to their anatomical and functional features. Bergmark developed a model by categorizing the "core" muscles as local and global. Local muscles provide stabilization between spinal segments, while global muscles are activated according to the direction of movement. The coordinated work of local and global muscles affects the quality of movements and "core" stability. "Core" muscles influence functional activities and functioning of the extremities by providing a stable basis for extremity movements and force transmission.

While core strength is defined as the muscular control mechanism that ensures functional stabilization of the spinal column, core endurance refers to the continuity of this control. Core endurance, a component of core stabilization, occurs when the lumbo-pelvic-hip muscles perform core contraction for a certain period of time or repeatedly. Although core strength plays a role by increasing internal-abdominal pressure to create resistance, core endurance allows muscles and muscle groups to remain in a stable position for a certain period of time. According to Lehman, core endurance affects spinal stabilization more than muscular strength due to the capacity of local core muscles to stabilize the lumbar spine. The "core" region functions as a connection point between the upper and lower extremities and enables the transfer of force from this region to the extremities. This region is a basic structure where the force required for all movements is generated and transmitted from the proximal segments to the distal segments.

During childhood and adolescence, physical and physiological changes vary suddenly depending on age and gender and last between the ages of 15-17. After the age of 18, change becomes regulated and physiological and performance values reach their maximum between the ages of 20-30. After the age of 30, functional capacity and other physical-physiological characteristics begin to decrease. The most important of these changes is the change in the skeletal-muscular system. Muscles develop from birth and reach their maximum level at the age of 25-30. As age progresses, the strength and cross-sections of muscle groups decrease. This decrease occurs faster in people who live sedentary lives.

The upper extremity is the primary tool humans use to manipulate the environment and has a wide range of capabilities with the same basic anatomical structures as the arm, forearm, hand, and fingers. In the upper extremity, mobility is more important than stability, and therefore the coordinated interaction of the shoulder complex, the functional unit of the upper extremity that enables movement relative to the trunk, provides sufficient stability despite high degrees of mobility. The primary function of the shoulder complex is to position the upper extremity so that the hand can function. The primary role of the elbow joint is to shorten or lengthen the length of the upper extremity. The hand is the structure responsible for performing the functions of the upper extremity and can perform many different activities as a manipulator and a means of communication. These activities require various characteristics such as positioning, strength, and precision, increasing their structural complexity compared to other joints of the upper extremity. However, there is a remarkable degree of synergy between these structures.

Reaction is the process by which an organism perceives and responds to stimuli. This process includes the stages in which muscles transmit impulses to the central nervous system (CNS) via afferent nerves, after the CNS decides which response to give, it sends this information back to the muscles via efferent nerves, and the muscles take action based on this information. Reaction time refers to the time between the moment a stimulus reaches the organism and the organism's response to this stimulus. Reaction time refers to the time it takes for an organism to respond to a particular stimulus and is generally divided into two main categories: simple and complex (complex) reaction time. Simple reaction time refers to the process of responding to a single stimulus. It can affect important physical parameters such as core endurance, upper extremity muscle strength, function and reaction time. However, there are not enough studies in the literature investigating this effect in healthy young adults. Most existing studies focus on the role of core endurance on athlete performance. The relationship between core endurance levels and upper extremity muscle strength, function and reaction time in healthy young adults has not yet been examined. The aim of our research is to examine the effect of core endurance levels on upper extremity function, muscle strength and reaction time in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-25.
* Individuals who volunteer to participate in the research.
* Individuals with normal joint movement.

Exclusion Criteria:

* Individuals with orthopedic or neurological diseases.
* Individuals who have suffered fractures, dislocations, surgeries, etc. in the upper extremities.
* Individuals with diseases that may affect upper extremity performance
* Individuals who exercise regularly
* Individuals who play any musical instrument

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 104 Healthy young adults
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Side bridge test | Day 1
  It is used to evaluate the endurance of the muscles (especially the obliques) located on the lateral side of the body. The individual lies sideways on the dominant side. When he is ready, he lifts his hips and stands on his forearm as long as he can, with his body in a single line, without any command. He puts his free hand on the opposite shoulder. The time period during which the position is maintained is recorded in seconds.
Prone bridge test (plank) test | Day 1
  It is used to evaluate the endurance of all core stabilization muscles together. The individual lies face down on his knees and forearms. When he is ready, he raises his knees so they are parallel to the ground and stands on his forearms and fingertips, without commands. The time it maintains the position is recorded in seconds.
Trunk flexion endurance test | Day 1
  It is used to evaluate the endurance of the trunk flexors, especially the abdominal muscles. The individual is in a supine position. When he is ready, he pulls his knees to his stomach so that they are parallel to the ground, without any command, and at the same time, with his arms tied, he lifts his upper body so that the lower end of the scapula lifts off the ground. The time it can maintain the position is recorded in seconds.
Sorensen test | Day 1
  It is used to evaluate the endurance of the back extensors. The individual lies face down on a stretcher high off the ground, with the upper body hanging off the bed. The individual's body part that comes into contact with the bed is positioned so that the anterior superior iliac spine is located. He maintains his balance with the help of a chair with his hands. The physiotherapist stabilizes the patient's legs. When the individual is ready, he crosses both hands on his shoulders and takes a position parallel to the ground, without taking any commands. The time it can maintain the position is recorded in seconds.

SECONDARY OUTCOMES:
Purdue Pegboard test | Day 1
  The Purdue Pegboard Test (PPT) is a test developed by J. Tiffin at Purdue University in 1948 to measure gross and fine motor skills of the hand, fingers, and arm. For the test, a test board with dimensions of 58.5x 29x 2.2 cm, 50 nails, 40 metal washers, small pipes through which the nails can pass and a stopwatch are used. The test board has four compartments and holes to insert the nails. The test consists of four subtests: Right hand, left hand, two hands and two hand team building. In each subtest, nails are placed into the holes within 30 seconds, starting with the dominant hand. In the last subtest, nails, washers and rings are placed as a set with both hands within 1 minute.
Isometric hand dynamometer for muscle strength | Day 1
  A digital dynamometer will be used to measure muscle strength. Individuals are placed in standard positions and the dynamometer will be placed at standard points. Individuals will be asked to show maximum resistance against the dynamometer. For this purpose, a trial application will be made first. A 1-minute rest period will be given after each measurement. Measurements will be repeated 3 times and the highest value will be recorded. Measurements will be made for shoulder flexion and shoulder abduction muscle strength in both upper extremities. The average of the measurements will be used as data. To evaluate shoulder flexion muscle strength, the patient lies in a sitting position on a chair, with the shoulder in 90° flexion, the elbow and wrist in neutral, and the forearm in pronation. To assess shoulder abduction, the patient sits on the examination table or chair and the arm is held in 90° abduction from the body midline.
Nelson hand reaction test | Day 1
  Nelson hand reaction test is a test that measures hand reaction time using a ruler. In the test, the participant sits and holds his hand on the table and spreads his fingers 8-10 centimeters away from the table, with his thumb and index fingers parallel. The tester holds the ruler at the level of the participant's thumb and index finger and asks the participant to look at the middle of the ruler. When ready, he puts the ruler down and asks the participant to catch the ruler. The point where the ruler is captured indicates the participant's reaction time. The test is repeated five times and the two highest and lowest values are subtracted. Reaction time is calculated by taking the average of the remaining three values.

CONTACTS AND LOCATIONS:
Overall Officials: Agabek ORUNBAYEV Msc, Study Chair — Karabuk University; Feruza JUMAYEVA Physiotherapist, Study Chair — Karabuk University; Musa GÜNEŞ Msc, Study Director — Karabuk University; Metehan YANA PhD, Principal Investigator — Karabuk Univeristy
Locations (1):
- Karabuk University, Karabük, Turkey (Türkiye)

REFERENCES:
- [Background] Bliss LS, Teeple P. Core stability: the centerpiece of any training program. Curr Sports Med Rep. 2005 Jun;4(3):179-83. doi: 10.1007/s11932-005-0064-y. PMID 15907272
- [Background] TIFFIN J, ASHER EJ. The Purdue pegboard; norms and studies of reliability and validity. J Appl Psychol. 1948 Jun;32(3):234-47. doi: 10.1037/h0061266. No abstract available. PMID 18867059
- [Background] Moreau CE, Green BN, Johnson CD, Moreau SR. Isometric back extension endurance tests: a review of the literature. J Manipulative Physiol Ther. 2001 Feb;24(2):110-22. doi: 10.1067/mmt.2001.112563. PMID 11208223
- [Background] Kibler WB, Press J, Sciascia A. The role of core stability in athletic function. Sports Med. 2006;36(3):189-98. doi: 10.2165/00007256-200636030-00001. PMID 16526831